CLINICAL TRIAL: NCT04616547
Title: A Single Arm Phase II Study of Bone-Targeted Sn-117m-DTPA in Symptomatic Castration Resistant Prostate Cancer With Skeletal Metastases
Brief Title: Treatment of Cancer-Related Bone Pain by Using Bone-Targeted Radiation-Based Therapy (Sn-117m-DTPA) in Patients With Prostate Cancer That Has Spread to Bones
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient drug supply
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2020-08371; NCI-2020-08371 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10437 (Other: Ohio State University Comprehensive Cancer Center LAO); 10437 (Other: CTEP); UM1CA186712 (NIH)
Record Dates: First submitted 2020-11-04; First posted 2020-11-05 (Actual); Results first posted 2024-04-16 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Castration-Resistant Prostate Carcinoma; Metastatic Malignant Neoplasm in the Bone; Metastatic Prostate Adenocarcinoma; Stage IV Prostate Cancer AJCC v8; Stage IVA Prostate Cancer AJCC v8; Stage IVB Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Pentetic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tin Sn 117m DTPA (Experimental): Patients receive tin Sn 117m DTPA IV over 5-10 minutes on day 1. Treatment repeats every 8 weeks for 2 cycles in the absence of disease progression or unacceptable toxicity. Patients may receive tin Sn 117m DTPA for an additional 2 cycles if pain recurs within 6 months after a 16-week pain observation period and no disease progression on bone scans, or evidence of clinical progression.
  Interventions: Other: Questionnaire Administration; Radiation: Tin Sn 117m Pentetate

INTERVENTIONS:
Other: Questionnaire Administration — Ancillary studies
Radiation: Tin Sn 117m Pentetate — Given IV
  Other Names: PENTETATE STANNIC SN-117M; Sn 117m Pentetic Acid; Sn-117m DTPA; Tin Sn 117m DTPA

SUMMARY:
This phase II trial studies the effect of Sn-117m-DTPA on bone pain in patients with prostate cancer that has spread to the bones. Sn-117m-DTPA is a radioactive therapeutic agent that localizes to bones when given to patients. Sn-117m-DTPA may help reduce bone pain in patients with prostate cancer that has spread to the bones.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the efficacy of tin-117m diethylenetriaminepentaacetic acid (Sn-117m-DTPA) on sustained pain response in patients with castration-resistant prostate cancer (CRPC) metastatic to at least two bone sites with at least one clinically meaningful pain at baseline (>= 4 on an 11-point pain intensity scale).

SECONDARY OBJECTIVES:

I. To assess the safety and tolerability of Sn-117m-DTPA per Common Terminology Criteria for Adverse Events (CTCAE) version (v)5.0.

II. To measure Sn-117m-DTPA activity by gamma-camera dosimetry scans (serial full body planar images) obtained at 1 hour, 4 hours (or within 4-6 hours), 24 hours (or within 16-24 hours), 48 hours (or within 36-48 hours), 72 hours (or within 60-72 hours), 1 week (+/- 2 days), and 4 weeks (+/- 2 days) after the first Sn-117m-DTPA administration.

III. To evaluate the therapeutic efficacy of Sn-117m-DTPA at 24 weeks as measured by Prostate Cancer Working Group 3 (PCWG3) criteria.

IV. To evaluate time to the first symptomatic skeletal event defined as i) the first use of external-beam radiation therapy to relieve skeletal symptoms; ii) new symptomatic pathologic vertebral or nonvertebral bone fractures; iii) spinal cord compression; or iv) tumor-related orthopedic surgical intervention.

V. To evaluate the overall pain response rate at 24 weeks. VI. To evaluate the duration of pain response defined as from the time of improvement in pain response (pain index =< 3) until the pain recurs.

VII. To measure changes and time to progression in serum prostate-specific antigen (PSA) and serum alkaline phosphatase (ALP) levels.

VIII. To measure patient-reported outcomes (PROs) and adverse events (AEs) (PRO-CTCAE) captured by digital instruments.

IX. To evaluate progression-free survival (PFS) and overall survival (OS).

EXPLORATORY OBJECTIVES:

I. To examine any tumor genomic alterations that may be associated with response or resistance to Sn-117m-DTPA, a radiopharmaceutical agent.

II. To examine the changes in systemic inflammatory markers (such as interferon [IFN]-gamma, tumor necrosis factor [TNF]-alpha, interleukins [IL]-8, IL-10, and IL-17) by flow cytometry, and changes in markers of immune function by measuring the percentage and absolute number of CD4+ T helper cells, CD8+ T cytotoxic cells, T regulatory cells, polymorphonuclear (PMN) myeloid-derived suppressor cells (MDSCs), and mononuclear MDSCs (M-MDSCs) prior to treatment versus (vs.) end of cycle 1, end of cycle 2, and at week 24 and correlate values and/or changes with treatment outcomes.

III. To evaluate the feasibility of measuring polo-like kinase 1 (Plk1) expression via immunohistochemistry (IHC) staining on archival tissues.

OUTLINE:

Patients receive tin Sn 117m DTPA intravenously (IV) over 5-10 minutes on day 1. Treatment repeats every 8 weeks for 2 cycles in the absence of disease progression or unacceptable toxicity. Patients may receive tin Sn 117m DTPA for an additional 2 cycles if pain recurs within 6 months after a 16-week pain observation period and no disease progression on bone scans, or evidence of clinical progression.

After completion of study, patients are followed up every 4 weeks until week 28, and then every 3 months for up to 12 months after the first dose of tin Sn 117m DTPA.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed adenocarcinoma of the prostate that is castration-resistant, defined as:

  * A castrate serum testosterone level =< 50 ng/dL or 1.7 nmol/L
  * Bilateral orchiectomy or maintenance on androgen ablation therapy with luteinizing hormone-releasing hormone (LHRH). Androgen deprivation therapy needs to be maintained throughout the study unless a patient has had orchiectomy by surgery
  * Serum PSA progression defined as two consecutive increases in PSA over a previous reference value, each measurement at least 1 week apart
* Progression after androgen receptor blockers (enzalutamide, apalutamide, or darolutamide) or androgen synthesis blockers (abiraterone acetate) or chemotherapy (docetaxel or cabazitaxel). There are no maximum number of prior therapies
* Progressive castration-resistant prostate cancer with two or more skeletal metastases identified by Tc-99m bone scintigraphy or prostate specific membrane antigen (PSMA) positron emission tomography (PET) scan
* Patients must have self-reported moderate to severe pain at trial entry (baseline weekly average "worst pain in the past 24-hours" scores of >= 4 on an 11-point numeric rating scale [NRS], the Brief Pain Inventory - Short Form [BPI-SF] item #3 for worst pain)
* Patients must either currently employ regular (not occasional) analgesic medication use for cancer-related bone pain or have undergone treatment with external beam radiation therapy (EBRT) for bone pain within 4 weeks before starting study treatment
* Age >= 18 years. Children < 18 years of age are excluded from the study as the prevalence of prostate cancer is extremely rare in this age group
* Patients must have a life expectancy >= 3 months
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Patients must have a serum PSA value >= 1 ng/mL
* Absolute neutrophil count >= 1,000/mcL
* Platelets >= 100,000/mcL
* Hemoglobin > 10.0 g/dL
* Total bilirubin =< 2.5 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT)(serum glutamic pyruvic transaminase [SGPT]) =< 5 x institutional ULN
* Creatinine =< 1.7 mg/dL OR glomerular filtration rate (GFR) >= 50 mL/min/1.73 m^2
* Patients receiving bisphosphonates prior to enrollment can maintain bisphosphonate therapy throughout all or part of the study. The bisphosphonate may be stopped or started at the discretion of the investigator throughout the study (i.e., both treatment phase and follow-up). Injection of bisphosphonates should be done at least 2 hours before or after study drug administration
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association functional classification. To be eligible for this trial, patients should be class 2B or better
* The effects of Sn-117m-DTPA on the developing human fetus are unknown. For this reason and because radionuclides are known to be teratogenic, male participants and their female partners must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while her male partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 6 months after completion of Sn-117m-DTPA administration
* Patients must be willing and able to comply with the protocol and agree to return to the hospital for follow-up visits and examinations
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients must not have visceral metastases (such as liver and lung) as assessed by abdominal/pelvic computed tomography (CT) or chest X-ray within 12 weeks before starting study treatment
* Patients must not have malignant lymphadenopathy exceeding 3 cm in short-axis diameter
* Patients must not have imminent or established spinal cord compression based on clinical findings and/or magnetic resonance imaging (MRI)
* Patients who have had chemotherapy, immunotherapy, or external radiotherapy within 4 weeks prior to entering the study
* Patients must not have received systemic radiotherapy with radium-223, strontium-89, samarium-153, rhenium-186, or rhenium-188 for the treatment of bony metastases within 24 weeks before starting study treatment
* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1) with the exception of alopecia
* Patients must not have received any investigational agents within 4 weeks before starting study treatment, nor be scheduled to receive one during the planned treatment period
* Patients must not have unmanageable urinary incontinence
* Patients must not have had known non-pathological bone fractures within 2 months before starting study treatment
* Patients must not have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to Sn-117m-DTPA
* Patients must not have uncontrolled intercurrent illness, including:

  * Any uncontrolled infection
  * Grade 2 or greater motor or sensory neuropathy
  * Crohn's disease or ulcerative colitis
* Patients with psychiatric illness/social situations that would limit compliance with study requirements

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-12-18 (Actual); Primary Completion 2022-02-16 (Actual); Study Completion 2022-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zin W Myint, Principal Investigator — Ohio State University Comprehensive Cancer Center LAO
Locations (1):
- University of Kentucky/Markey Cancer Center, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

REFERENCES:
- [Derived] Myint ZW, El Khouli R, Lemieux B, Yan D, St Clair WH, Liu X, Kunos CA. A single arm phase II study of bone-targeted Sn-117 m-DTPA in symptomatic castration-resistant prostate cancer with skeletal metastases. BMC Cancer. 2022 Apr 15;22(1):415. doi: 10.1186/s12885-022-09496-2. PMID 35428207

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tin Sn 117m DTPA
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Tin Sn 117m DTPA
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Sustained Pain Response
Description: Defined as achieving pain index =< 3 within a 12-week period, maintaining that pain index =< 3 over a 16-week time period. Will also be summarized by the point estimation of the overall response rate (ORR) with the corresponding 95% confidence intervals. Patients who received any amount of study drug will be included in the denominator for the calculation of ORR.
Time Frame: Baseline to 16 weeks
Population: Data not collected and analyzed due to low enrollment to the study
Arm/Group | Tin Sn 117m DTPA
Number analyzed (Participants) | 0

2. Secondary Outcome: Incidence of Adverse Events (AEs)
Description: Safety and toxicity will be assessed through the frequency and percent of AEs, serious adverse events, and adverse events of special interests. Toxicity will be assessed using Common Terminology Criteria for Adverse Events. Will be assessed by patient reported outcomes (PROs) and AEs (PRO-Common Terminology Criteria for Adverse Events).
Time Frame: Up to 6 months post-therapy
Population: Data not collected and analyzed due to low enrollment to the study
Arm/Group | Tin Sn 117m DTPA
Number analyzed (Participants) | 0

3. Secondary Outcome: Tin Sn 117m Diethylenetriaminepentaacetic Acid (DTPA) (Sn-117m-DTPA) Activity
Description: Gamma camera dosimetry will be used to evaluate whole-body distribution of Sn-117m-DTPA. Pearson's correlation coefficient method will be used to assess the correlation between the baseline technetium-99 bone scintigraphy measurement and the Sn-117m-DTPA uptake. If the observed data distribution is not appropriate to calculate the Pearson's correlation, post hoc analysis will be conducted using non-parametric methods or other methods suitable to the observed data distribution. The gamma dosimetry scan measurements will be reported descriptively as the average and standard deviation of dosimetry scan measurements and plotted over time and grouped by organ systems.
Time Frame: Up to 4 weeks after the first Sn-117m-DTPA administration
Population: Data not collected due to low enrollment to the study
Arm/Group | Tin Sn 117m DTPA
Number analyzed (Participants) | 0

4. Secondary Outcome: Overall Response Rate
Description: A Fisher's exact 95% confidence interval will be calculated for the overall response rate. The denominator will include all patients who received at least one dose of study treatment and do not have major protocol deviations. Patients who do not have observed clinical response will be counted as negative responses.
Time Frame: Up to 12 months after the first dose of tin Sn 117m DTPA
Population: Data not collected and analyzed due to low enrollment to the study
Arm/Group | Tin Sn 117m DTPA
Number analyzed (Participants) | 0

5. Secondary Outcome: Time to First Symptomatic Skeletal Event
Description: The time from study enrollment to the first use of external-beam radiation therapy to relieve skeletal symptoms, new symptomatic pathologic vertebral or non-vertebral bone fractures, spinal cord compression, or tumor-related orthopedic surgical intervention will be evaluated. Will be analyzed using the Kaplan-Meier method. Estimation and confidence intervals for the median time to first symptomatic skeletal event will be provided.
Time Frame: Up to 12 months
Population: Data not collected and analyzed due to low enrollment to the study
Arm/Group | Tin Sn 117m DTPA
Number analyzed (Participants) | 0

6. Secondary Outcome: Overall Pain Response Rate
Description: The rate of achievement of pain index =< 3 within 12 weeks from the first Sn-117m-DTPA will be evaluated.
Time Frame: Within 12 weeks from first dose of Sn-117m-DTPA
Population: Data not collected and analyzed due to low enrollment to the study
Arm/Group | Tin Sn 117m DTPA
Number analyzed (Participants) | 0

7. Secondary Outcome: Duration of Pain Response
Time Frame: Time from the achievement of pain response (pain index =< 3) to the recurrence of pain (pain index >= 4), assessed up to 16 weeks
Population: Data not collected and analyzed due to low enrollment to the study
Arm/Group | Tin Sn 117m DTPA
Number analyzed (Participants) | 0

8. Secondary Outcome: Prostate Specific Antigen (PSA) Response Rates
Description: Will be determined for the following benchmarks: >= 30% reduction of the blood level, compared to the baseline value; >= 50% reduction of the blood level, compared to the baseline value; confirmed PSA response: >=50% reduction of the blood level, compared to the baseline value, and confirmed by a second PSA value approximately 4 or more weeks later.
Time Frame: Up to 28 weeks
Population: Data not collected and analyzed due to low enrollment to the study
Arm/Group | Tin Sn 117m DTPA
Number analyzed (Participants) | 0

9. Secondary Outcome: Alkaline Phosphatase (ALP) Response Rate
Description: Will be determined for the following benchmarks: >= 50% reduction of the blood level, compared to the baseline value; confirmed ALP response: >= 50% reduction of the blood level, compared to the baseline value, and confirmed by a second ALP value approximately 4 or more weeks later.
Time Frame: Up to 28 weeks
Population: Data not collected and analyzed due to low enrollment to the study
Arm/Group | Tin Sn 117m DTPA
Number analyzed (Participants) | 0

10. Secondary Outcome: Clinical Progression-free Survival
Description: Defined as symptomatic progression (increasing pain from a metastatic lesion); progression of bone lesions assessed per Prostate Cancer Working Group 3 criteria; or progression of soft-tissue lesions assessed per Response Evaluation Criteria in Solid Tumors version 1.1 criteria. PSA progression without progression on bone lesions nor symptomatic is not considered as clinical progression. Will be summarized by Kaplan-Meier methods.
Time Frame: Time of study enrollment until disease progression, assessed up to 12 months
Population: Data not collected and analyzed due to low enrollment to the study
Arm/Group | Tin Sn 117m DTPA
Number analyzed (Participants) | 0

11. Secondary Outcome: Overall Survival
Description: Will be summarized by Kaplan-Meier methods.
Time Frame: Time of the first study treatment until the date of death, assessed up to 12 months
Population: Data not collected and analyzed due to low enrollment to the study
Arm/Group | Tin Sn 117m DTPA
Number analyzed (Participants) | 0

12. Other Pre Specified Outcome: Tumor Genomic Alterations
Time Frame: Up to 12 months
Population: Data not collected and analyzed due to low enrollment to the study
Arm/Group | Tin Sn 117m DTPA
Number analyzed (Participants) | 0

13. Other Pre Specified Outcome: Changes in Systemic Inflammatory Markers and Immune Cell Populations
Description: Will be summarized using descriptive statistics.
Time Frame: Baseline to after completion of treatment
Population: Data not collected and analyzed due to low enrollment to the study
Arm/Group | Tin Sn 117m DTPA
Number analyzed (Participants) | 0

14. Other Pre Specified Outcome: Polo-like Kinase 1 Immunohistochemistry
Description: Will be summarized using descriptive statistics.
Time Frame: Up to 12 months
Population: Data not collected and analyzed due to low enrollment to the study
Arm/Group | Tin Sn 117m DTPA
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: The NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 was used for grading patients adverse events. Adverse events were collected and monitored from the start of the study until study completion up to an average of 6 months.
Arm/Group | Tin Sn 117m DTPA
All-Cause Mortality (participants affected / at risk) | 1/1
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tin Sn 117m DTPA (N=1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Skin Infection (Skin and subcutaneous tissue disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tin Sn 117m DTPA (N=1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dysphasia (Nervous system disorders) | 1 (1)
Ear and Labyrinth (Ear and labyrinth disorders) | 1 (1) — Cerumen Impaction
Edema limbs (General disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Injection site reaction (Injury, poisoning and procedural complications) | 1 (1)
Lymphocyte count increased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Weight loss (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-10): https://cdn.clinicaltrials.gov/large-docs/47/NCT04616547/Prot_SAP_000.pdf
  • Informed Consent Form (2022-01-10): https://cdn.clinicaltrials.gov/large-docs/47/NCT04616547/ICF_001.pdf